CLINICAL TRIAL: NCT05776524
Title: A Phase 2 Study of Amplitude-Modulated Radiofrequency Electromagnetic Fields in Metastatic Pancreatic Cancer
Brief Title: Study of Amplitude-Modulated Radiofrequency Electromagnetic Fields in Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: THERABIONIC INC. (Other)
Collaborators: Therabionics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094460; WFBCCC 57122 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer; Metastatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Taxes; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- GEM-ABR [Gemcitabine - Abraxane (nab-Paclitaxel)] with TheraBionic device (Experimental): Metastatic pancreatic cancer patients will be treated with amplitude-modulated radiofrequency electromagnetic fields using TheraBionic device in combination with standard chemotherapy, gemcitabine- nab-paclitaxel. amplitude-modulated radiofrequency electromagnetic fields will be delivered by the TheraBionic device.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Device: TheraBionic

INTERVENTIONS:
Drug: Nab paclitaxel — 125 mg/m2 weekly, on days 1,8, and 15 or on days 1 and 15 as a 30-40 minute infusion administered first
Drug: Gemcitabine — 1000 mg/m2 weekly, on day 1,8 and 15 or 1000 mg/m2 weekly, on day 1 and 15 over 30 minutes after nab- paclitaxel infusion
Device: TheraBionic — This treatment consists of delivering low levels of radio waves into the body with a spoon-shaped antenna placed in the mouth, three times a day, for an hour each time.

SUMMARY:
The objective of this research is to find out what effects (good and bad), the combination of gemcitabine and nab-paclitaxel therapy (GEM-ABR for the rest of the document), standard chemotherapy for pancreatic cancer, and the TheraBionic device has on participants' condition.

DETAILED DESCRIPTION:
Primary Objective(s): The primary objective of this study is to evaluate the efficacy of the combination of nab-paclitaxel, gemcitabine, and amplitude-modulated radiofrequency electromagnetic fields in improving 6-month overall survival (OS) rates in patients with metastatic adenocarcinoma of the pancreas.

Secondary Objective(s):

* Evaluate the safety and tolerability of the combination of nab-paclitaxel, gemcitabine, and amplitude-modulated radiofrequency electromagnetic fields in patients with metastatic adenocarcinoma of the pancreas.
* Evaluate progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) guidelines in patients with metastatic adenocarcinoma of the pancreas treated with the combination of nab-paclitaxel, gemcitabine, and amplitude-modulated radiofrequency electromagnetic fields.
* Evaluate the objective response rate (ORR) in patients with metastatic adenocarcinoma of the pancreas treated with the combination of nab-paclitaxel, gemcitabine, and amplitude-modulated radiofrequency electromagnetic fields.
* Evaluate the disease control rate (DCR) in patients with metastatic adenocarcinoma of the pancreas treated with the combination of nab-paclitaxel, gemcitabine, and amplitude-modulated radiofrequency electromagnetic fields.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have newly diagnosed untreated biopsy proven metastatic adenocarcinoma of the pancreas. If a patient had a biopsy of the pancreatic mass and the clinical picture is consistent with metastatic pancreatic cancer, another biopsy of a metastatic site is not required for this trial. Pancreatic tumors with mixed histology that has predominant adenocarcinoma can be enrolled.
* One or more measurable metastatic tumors per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) on imaging studies (CT or MRI) of chest, abdomen and pelvis.
* Females of childbearing potential and males with female partners of childbearing potential, if sexually active, must agree to use two forms of contraception during the period of administration of study drug and up to 6 months after the end of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Age 18 years old or greater.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Patients must have organ and marrow function as defined below:

Organ and Marrow Function Absolute neutrophil count (ANC) ≥ 1,500/mcL Platelets* ≥ 100,000/mcL Hemoglobin* ≥ 7 g/dL *It is acceptable to transfuse packed red blood cells (PRBC) and platelets at the time of enrollment to meet the eligibility criteria.

Total bilirubin ≤ 1.5 X institutional upper limit of normal AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal (≤ 5 x ULN, if liver metastasis) Creatinine ≤ 1.5 X institutional upper limit of normal Or CrCL > 50

- Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Patients treated with any chemotherapy in metastatic setting and/or who had chemotherapy with gemcitabine and/or nab-paclitaxel within six months prior to entering the study in the adjuvant or neo-adjuvant setting are excluded. Patients who have had chemotherapy with FOLFIRINOX prior to entering the study in the adjuvant or neo-adjuvant setting can be enrolled into the study.
* Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine and nab-paclitaxel.
* History of malignancy in last 3 years except cervical cancer in situ, adequately treated basal cell or squamous cell carcinoma of skin or treated low risk prostate cancer, who are considered to be eligible.
* Patients receiving calcium channel blockers and any agent blocking L-type of T type Voltage Gated Calcium Channels such as amlodipine, nifedipine, ethosuximide are not allowed in the study unless their medical treatment is modified to exclude calcium channel blockers prior to enrollment.
* Patients with active and uncontrolled bacterial, viral or fungal infection requiring systemic therapy. Patients can be reevaluated for the study if the infection is deemed to be under control and the systemic therapy is completed.
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or could compromise patient safety.
* Known diagnosis of interstitial lung disease, sarcoidosis, pulmonary fibrosis or pneumonitis.
* Pregnant women are excluded from this study because of potential risk for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy and amplitude-modulated radiofrequency electromagnetic fields, patients who are breastfeeding will be excluded to participate in this study.
* Localized resectable or locally advanced tumor.
* Undergone surgery, other than diagnostic surgery or minor procedures, within 4 weeks prior to the treatment day.
* Unable to comply with study procedures or anticipating a situation that would result in a treatment break for 14 or more consecutive days after the start of the study.
* Actively enrolled in any other clinical interventional trial or receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | At 6 months
  Overall survival is defined from the time of study treatment initiation until death of any cause. Six months overall survival (OS 6) is defined as the proportion of patients alive at six months from treatment initiation. All participant demographic and clinical characteristics will be summarized using mean (standard deviation) and count (percent) for continuous and categorical variables, respectively. Primary analysis will calculate the overall survival rate at 6-months with one-sided 95% confidence interval

SECONDARY OUTCOMES:
Incidences of Adverse Events | Up to 1 year after treatment intervention
  The incidence of treatment-emergent toxicities/adverse events (AEs) and severe adverse events in terms categorized and graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5)
Progression-Free Survival | Up to 1 year
  Progression-free survival is defined from the time of study treatment (amplitude-modulated radiofrequency electromagnetic fields plus chemo) initiation until progression according to RECISTv1.1 guidelines or death of any cause, whichever occurs first, as measured throughout the study. Kaplan-Meier curves will be constructed to assess progression-free survival with estimated 6-month and median times with 95% confidence intervals
Tumor Response | Up to 1 year
  Objective tumor response based on CT or MRI scans. These will be evaluated according to the RECISTv1.1 criteria:
  1. Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 2.0 cm by chest x-ray, by ≥ 1.0 cm with CT or MRI scans, or ≥ 1.0 cm with calipers by clinical exam.
  2. Malignant lymph nodes are to be considered pathologically enlarged and measurable if it measures ≥ 1.5 cm in short axis (greatest diameter perpendicular to the long axis of the lymph node) when assessed by scan (CT scan slice recommended being no greater than 0.5 cm).
  Tumor response will be summarized by count/percent with one-sided Clopper Pearson exact 95% confidence interval.
Disease Control Rate | Up to 1 year
  Disease control rate defined as the proportion of patients with disease control (complete or partial response or stable disease) based on RECISTv1.1 criteria:
  1. Complete Response (CR): Complete disappearance of all target and non-target lesions. No new lesions. No disease related symptoms. Any lymph nodes must have reduction in short axis to < 1.0 cm.
  2. Partial Response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
  3. Stable Disease (SD): Does not qualify for CR, PR, Progression or Symptomatic Deterioration.
  Disease control rate will be summarized by count/percent with one-sided Clopper Pearson exact 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Paluri, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No